CLINICAL TRIAL: NCT02754089
Title: The Effects of Rhus Coriaria L. (Rhus or Somagh) on Body Weight
Brief Title: The Effects of Rhus Coriaria L. on Body Weight
Acronym: SomaghWeight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mesbah Shams, MD, Associate professor of Internal Medicine & Endocrinology, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-92-5581
Record Dates: First submitted 2016-04-26; First posted 2016-04-28 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2016-09

CONDITIONS: Body Weight
Keywords: Body weight changes; Medicine, Traditional; Herbal medicine; Rhus; Waist Circumference; Waist-Hip Ratio; Body mass index
MeSH Terms: conditions — Body Weight; Body Weight Changes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rhus (Experimental): 500 mg twice daily after meal for 6 weeks
  Interventions: Drug: Rhus Coriaria L.(Rhus)
- Placebo (Placebo Comparator): 500 mg twice daily after meal for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rhus Coriaria L.(Rhus) — 500 mg twice daily after meals for 6 weeks
  Other Names: Somagh
  Arms: Rhus
Drug: Placebo — 500 mg twice daily after meals for 6 weeks
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the effects of Rhus coriaria L. (Rhus) commonly known as "Somagh" on body weight.

DETAILED DESCRIPTION:
Rhus coriaria L.(Rhus) is a well-known spice widely consumed in the world which has also been utilized extensively for medicinal purposes. The antioxidant components of this plant made it a favorable target for laboratory and animal studies in different conditions such as oxidative stress cytotoxicity, diabetes and hyperlipidemia. Rhus (Somagh) is found in temperate and tropical regions worldwide, often growing in areas of marginal agricultural capacity. Rhus is used as an herbal remedy in traditional medicine because of its assumed analgesic, antidiarrheic, antiseptic, anorexic and antihyperglycemic properties. The fruits of Rhus contain flavonols, phenolic acids, hydrolysable tannins, anthocyans and organic acids such as malice, citric and tartaric acids. Some studies have shown that polyphenols could have beneficial effects on cardiovascular disease and cancer and could be regarded as bioactive compounds with a high potential health-promoting capacity. Phenolic compounds inhibit lipid peroxidation, scavenge the superoxide anion and hydroxyl radical, and enhance the activities of detoxifying enzymes.

The aim of this study is to evaluate the effects of Rhus coriaria L. (Rhus) commonly known as Somagh on body weight.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) >= 25 kg/m2

Exclusion Criteria:

* Diabetes mellitus
* Hypo. or hyperthyroidism
* Any systemic illnesses e.g. liver cirrhosis, acute or chronic renal failure, heart failure
* Use of drugs: Weight lowering agents, glucocorticoids, Oral contraceptive pills.
* Pregnancy
* History of allergic reaction to Somagh

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | 6 weeks

SECONDARY OUTCOMES:
Waist Circumference (cm) | 6 weeks
Hip Circumference (cm) | 6 weeks
Leptin (ng/ml) | 6 weeks
Insulin (mU/l) | 6 weeks
Fasting Blood Glucose (mg/dl) | 6 weeks
Number of patients with adverse event | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mojtaba Heydari, MD, Principal Investigator — Research Center for Traditional Medicine and History of Medicine, Shiraz University of Medical Sciences, Shiraz, IR Iran; Gholamhossein Ranjbar Omrani, MD, Study Chair — Endocrine and Metabolism Research Center, Shiraz University of Medical Sciences; Zahra Hajmohammadi, MD, Principal Investigator — Department of Internal Medicine, Shiraz University of Medical Sciences, Shiraz, Iran
Locations (1):
- Shahid Motahhari Clinic, Shiraz University of Medical Sciences, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: Undecided